CLINICAL TRIAL: NCT04104438
Title: A Study in Adults on Pre LT Dialysis With Basiliximab, Delayed Tacrolimus (TAC), Mycophenolate (MMF), Steroids (Grp 1) vs. Basiliximab, Delayed TAC, MMF, Steroids, With Everolimus 30d Post LT(Grp 2), vs. TAC, MMF, Steroids (Grp 3).
Brief Title: Examination of Immunosuppression Adjustment Impact on Kidney Function in Liver Transplant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fady M Kaldas, M.D., F.A.C.S. (Other)
Responsible Party: Sponsor-Investigator, Fady M Kaldas, M.D., F.A.C.S., Clincal Professor of Surgery, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Novartis18-000215
Record Dates: First submitted 2019-05-30; First posted 2019-09-26 (Actual); Results first posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Asses Immunosuppression Modulation on Renal Recovery Post LT
MeSH Terms: interventions — Basiliximab; Everolimus

STUDY DESIGN:
Intervention Model Description: To assess the efficacy and safety of basiliximab, delayed dose tacrolimus plus mycophenolate mofetil, and SOC corticosteroids versus basiliximab, delayed dose tacrolimus plus mycophenolate mofetil, and SOC corticosteroids and addition of delayed everolimus/mycophenolate minimization at one month post OLT compared to standard triple immunosuppression (tacrolimus, mycophenolate mofetil and corticosteroids) for prevention of acute organ rejection in liver transplant recipients with a high risk of developing renal dysfunction following OLT or with concomitant renal dysfunction prior to OLT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- basiliximab with Delayed TAC (Active Comparator): basiliximab
  * Dose #1: 20mg IV within 2 hours of transplant
  * Dose #2: 20mg IV Post-operative day #4
  Tacrolimus (with basiliximab induction) o Beginning day #5 post-transplant or when SCr < 1.8 mg/dl (subjects off dialysis) to six months: 0.03-0.1mg/kg q12h PO to maintain whole blood trough concentration of 4-6ng/mL
  Mycophenolate mofetil
  o 1000 mg po bid
  Corticosteroids (SOC): Per UCLA protocol
  Post-operative taper:
  * Post-op day 1- methylprednisolone 50mg IVP Q6H
  * Post-op day 2- methylprednisolone 40mg IVP Q6H
  * Post-op day 3- methylprednisolone 30mg IVP Q6H
  * Post-op day 4- methylprednisolone 20mg IVP Q6H
  * Post-op day 5- methylprednisolone 20mg IVP Q12H
  * Post-op day 6- methylprednisolone 10mg IVP Q12H until taking PO, then change to: prednisone 20mg PO QAM
  Interventions: Drug: Basiliximab 20 MG
- basiliximab, Delayed TAC with Everolimus (Active Comparator): basiliximab
  Tacrolimus (with basiliximab induction)
  o Beginning day #5 post-transplant or when SCr < 1.8 mg/dl (subjects off dialysis) to POD 30: 0.03-0.1mg/kg q12h PO to maintain whole blood trough concentration of 4-6ng/mL
  Mycophenolate mofetil o 1000 mg po bid up to POD 30: reduce mycophenolate mofetil following achievement of steady state everolimus (POD 35) as clinically indicated
  Corticosteroids (SOC): Per UCLA protocol
  Everolimus (delayed)
  o Add by POD 30: 1 mg po bid and adjusted to maintain whole blood trough concentrations of 3-8 ng/ml.
  Interventions: Drug: Basiliximab 20 MG
- Control: standard TAC with steroids and MMF (No Intervention): Tacrolimus (without basiliximab induction)
  * Beginning day #1 post-transplant to six months: 0.03-0.1mg/kg q12h po to maintain whole blood trough concentration of 5-12ng/mL
  * Six months to one year: maintain whole blood trough concentration of 5-10ng/mL
  Mycophenolate mofetil
  o 1000 mg po bid
  Corticosteroids (SOC): Per UCLA protocol

INTERVENTIONS:
Drug: Basiliximab 20 MG — Basiliximab induction followed by tacrolimus, corticosteroids and mycophenolic acid with a switch to everolimus by post operative day 30
  Other Names: Everolimus
  Arms: basiliximab with Delayed TAC; basiliximab, Delayed TAC with Everolimus

SUMMARY:
This is a study to help understand how well new combinations of immunosuppressive medications (medications that weaken your immune system to prevent your body from rejecting the transplanted liver) work compared to standard immunosuppressive medications after your liver transplant. Also the study will assess how safe the new combination of immunosuppressive medicines are and if there are any changes in how your kidneys work after taking these medicines.

DETAILED DESCRIPTION:
A single center, open label, randomized, prospective, pilot study of induction and maintenance immunosuppression in adult subjects >18 years undergoing orthotopic liver transplantation (OLT) with Basiliximab, delayed dose tacrolimus plus mycophenolate mofetil and standard of care (SOC) corticosteroids (Group 1) versus basiliximab, delayed dose tacrolimus plus mycophenolate mofetil, SOC corticosteroids, with addition of delayed maintenance Everolimus at one month post OLT with subsequent mycophenolate mofetil minimization (Group 2) versus standard dose tacrolimus plus mycophenolate mofetil plus SOC corticosteroids (Group 3; control) with concomitant renal dysfunction prior to OLT.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for inclusion in this study have to fulfill all of the following criteria:

  1. A signed informed consent prior to patient participation in the study and before any assessment is performed.
  2. Patients who are able to take oral medication.
  3. 18 years old
  4. Undergoing first OLT
  5. Dialysis for 45 days or less at time of transplant
  6. Able and willing to conform to requirements of the study
  7. Able and willing to provide informed consent

     Exclusion Criteria:

  <!-- -->

  1. < 18 years old
  2. Autoimmune liver disease, Primary Sclerosing Cholangitis, Primary Biliary Cirrhosis
  3. Dialysis greater than 45 days
  4. Receiving ATG, IVIG therapy, or sirolimus/everolimus around time of transplant or sirolimus/everolimus after transplant
  5. Unable to take oral medications
  6. Participating in another clinical research study involving the evaluation of another investigational drug or device
  7. Documented allergy to basiliximab, TAC, MMF or any macrolide antibiotic.
  8. Presence of thrombosis of any major hepatic arteries
  9. Complex/high risk arterial reconstruction at any time (graft vessel patency by Doppler ultrasound confirmed and documented).
  10. Patients who are recipients of multiple solid organ transplants, (e.g., multivisceral or combined liver-kidney transplants), or have previously received an organ or tissue transplanted, or who received an ABO incompatible transplant.
  11. Patients who have severe hypercholesterolemia (>215 mg/dL; >5.5 mmol/L) or hypertriglyceridemia (>265 mg/dL; >3.0 mmol/L) at Baseline.
  12. Patients who have severe thrombocytopenia or neutropenia (platelet count >20 and MLCs>1000)
  13. Patients who have any surgical or medical condition, which in the opinion of the investigator, might significantly alter the absorption, distribution, metabolism and excretion of study drugs
  14. Patients with a known hypersensitivity to the drugs used on study or their class, or to any of the excipients.
  15. Patients with clinically significant systemic infection
  16. Pregnant or nursing (lactating) female patients, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive βHCG laboratory test (>9 mIU/mL) at Baseline.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fady M Kaldas, MD, Principal Investigator — UCLA Dept Surgery
Locations (1):
- UCLA Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Basiliximab With Delayed TAC: Basiliximab
  * Dose #1: 20mg IV within 2 hours of transplant
  * Dose #2: 20mg IV Post-operative day #4
  Tacrolimus (with basiliximab induction) o Beginning day #5 post-transplant or when SCr < 1.8 mg/dl (subjects off dialysis) to six months: 0.03-0.1mg/kg q12h PO to maintain whole blood trough concentration of 4-6ng/mL
  Mycophenolate mofetil
  o 1000 mg po bid
  Corticosteroids (SOC): Per UCLA protocol
  Post-operative taper:
  * Post-op day 1- methylprednisolone 50mg IVP Q6H
  * Post-op day 2- methylprednisolone 40mg IVP Q6H
  * Post-op day 3- methylprednisolone 30mg IVP Q6H
  * Post-op day 4- methylprednisolone 20mg IVP Q6H
  * Post-op day 5- methylprednisolone 20mg IVP Q12H
  * Post-op day 6- methylprednisolone 10mg IVP Q12H until taking PO, then change to: prednisone 20mg PO QAM
  Basiliximab 20 MG: Basiliximab induction followed by tacrolimus, corticosteroids and mycophenolic acid with a switch to everolimus by post operative day 30
- Basliximab, Delayed TAC With Everolimus: Basiliximab
  Tacrolimus (with basiliximab induction)
  o Beginning day #5 post-transplant or when SCr < 1.8 mg/dl (subjects off dialysis) to POD 30: 0.03-0.1mg/kg q12h PO to maintain whole blood trough concentration of 4-6ng/mL
  Mycophenolate mofetil o 1000 mg po bid up to POD 30: reduce mycophenolate mofetil following achievement of steady state everolimus (POD 35) as clinically indicated
  Corticosteroids (SOC): Per UCLA protocol
  Everolimus (delayed)
  o Add by POD 30: 1 mg po bid and adjusted to maintain whole blood trough concentrations of 3-8 ng/ml.
  Basiliximab 20 MG: Basiliximab induction followed by tacrolimus, corticosteroids and mycophenolic acid with a switch to everolimus by post operative day 30
Period: Overall Study
Arm/Group | Basiliximab With Delayed TAC | Basliximab, Delayed TAC With Everolimus | Control: Standard TAC With Steroids and MMF
Started | 30 | 28 | 13
Completed | 28 | 20 | 11
Not Completed | 2 | 8 | 2
Not completed — Death | 2 | 1 | 2
Not completed — Adverse Event | 0 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Disenrolled due to noncompliance | 0 | 1 | 0
Not completed — stopped due to possible operation | 0 | 1 | 0
Not completed — everolimus not started due to bile duct injury | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Basiliximab With Delayed TAC | Basliximab, Delayed TAC With Everolimus | Control: Standard TAC With Steroids and MMF | Total
Number analyzed (Participants) | 30 | 28 | 13 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 23 | 10 | 55
  >=65 years | 8 | 5 | 3 | 16
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55 [36 to 65] | 55 [40 to 61] | 59 [46 to 65] | 56 [25 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 6 | 32
  Male | 17 | 15 | 7 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 18 | 7 | 45
  Not Hispanic or Latino | 9 | 10 | 6 | 25
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Other race | 20 | 18 | 8 | 46
  African American | 0 | 1 | 3 | 4
  Asian | 3 | 2 | 0 | 5
  Caucasian | 5 | 7 | 2 | 14
  More than 1 race | 2 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 30 | 28 | 13 | 71

OUTCOME MEASURES:

1. Primary Outcome: Participants Who Have Recovered Renal Function
Description: Assessment of dialysis independence (patients no longer requiring dialysis post LT)
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Basiliximab With Delayed TAC | Basliximab, Delayed TAC With Everolimus | Control: Standard TAC With Steroids and MMF
Number analyzed (Participants) | 28 | 20 | 11
Participants | 28 | 20 | 11

2. Other Pre Specified Outcome: Cumulative Allograft Rejection
Description: Liver biopsy-proven rejection
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Basiliximab With Delayed TAC | Basliximab, Delayed TAC With Everolimus | Control: Standard TAC With Steroids and MMF
Number analyzed (Participants) | 28 | 20 | 11
Participants | 2 | 3 | 2

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Basiliximab With Delayed TAC | Basliximab, Delayed TAC With Everolimus | Control: Standard TAC With Steroids and MMF
All-Cause Mortality (participants affected / at risk) | 2/30 | 1/28 | 2/13
Serious Adverse Events (participants affected / at risk) | 14/30 | 7/28 | 1/13
Other Adverse Events (participants affected / at risk) | 14/30 | 18/28 | 8/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Basiliximab With Delayed TAC (N=30) | Basliximab, Delayed TAC With Everolimus (N=28) | Control: Standard TAC With Steroids and MMF (N=13)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Nausea/Vomiting (General disorders) | 2 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 2 | 0 | 0
Weakness (General disorders) | 1 | 0 | 0
Fever (General disorders) | 3 | 3 | 0
UTI (Renal and urinary disorders) | 0 | 1 | 1
Hyperkalemia (Renal and urinary disorders) | 1 | 2 | 0
encepahlopathy (Hepatobiliary disorders) | 1 | 2 | 0
kidney stone (Renal and urinary disorders) | 1 | 0 | 0
dysphagia (General disorders) | 1 | 0 | 0
stroke (General disorders) | 1 | 0 | 0
bile duct stricture (Hepatobiliary disorders) | 0 | 0 | 1
pyothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Basiliximab With Delayed TAC (N=30) | Basliximab, Delayed TAC With Everolimus (N=28) | Control: Standard TAC With Steroids and MMF (N=13)
Indigestion (Gastrointestinal disorders) | 0 | 0 | 1
hand/wrist pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
chest pain (General disorders) | 1 | 0 | 1
wound healing delay (General disorders) | 0 | 0 | 1
hyperkalemia (Renal and urinary disorders) | 1 | 1 | 2
hypotension (General disorders) | 0 | 0 | 1
abdominal pain (General disorders) | 1 | 5 | 0
diarrhea (Gastrointestinal disorders) | 1 | 2 | 0
insomnia (General disorders) | 0 | 1 | 0
nausea (General disorders) | 1 | 3 | 0
back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Lower extremity edema (General disorders) | 0 | 1 | 0
fatigue (General disorders) | 1 | 3 | 0
sore throat (General disorders) | 0 | 1 | 0
anemia (General disorders) | 3 | 0 | 0
dizziness (General disorders) | 1 | 0 | 0
neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0
tingling (General disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2023-11-07): https://cdn.clinicaltrials.gov/large-docs/38/NCT04104438/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-03): https://cdn.clinicaltrials.gov/large-docs/38/NCT04104438/SAP_001.pdf
  • Informed Consent Form (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/38/NCT04104438/ICF_003.pdf